CLINICAL TRIAL: NCT00991627
Title: Pharmacological or Non-Pharmacological Management of Maternal Hypotension During Elective Cesarean Section Under Subarachnoid Anesthesia: a Randomized, Controlled Trial
Brief Title: Different Approaches to Maternal Hypotension During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Guido Fanelli, UO II Anestesia, Rianimazione e Terapia Antalgica, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANEST-OST-02
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Pregnancy; Cesarean Section; Anesthesia,Spinal; Hypotension
Keywords: Ephedrine; Adrenergic Agents; Central Nervous System Stimulants; Sympathomimetics; Vasoconstrictor Agents; Bupivacaine; Anesthetics, Local; Atropine; Adjuvants, Anesthesia; Anti-Arrhythmia Agents; Bronchodilator Agents; Muscarinic Antagonists; Mydriatics; Parasympatholytics; Morphine; Analgesics, Opioid; Narcotics; Ringer's Lactate; Isotonic Solutions; Hypotension; Blood pressure; Signs and Symptoms; Pregnancy; Anesthesia, Obstetrical; Inferior Vena Cava
MeSH Terms: conditions — Hypotension; Signs and Symptoms | interventions — Bupivacaine; Anesthetics, Local; Morphine; Ringer's Lactate; Ephedrine; Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacological (Active Comparator): Patients in this group will receive a basal infusion of ephedrine. Hypotension will be treated for a reduction in systolic blood pressure 20% below baseline values.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Lactated Ringer's solution; Drug: Ephedrine, continuous infusion; Drug: Ephedrine, bolus; Drug: Atropine
- Non-Pharmacological (Experimental): Patients in this group will undergo uterine lateral displacement through the use of a wedge-shaped cushion placed under their right hip. Hypotension will be treated for a reduction in systolic blood pressure 40% below baseline values.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Lactated Ringer's solution; Drug: Ephedrine, bolus; Drug: Atropine

INTERVENTIONS:
Drug: Bupivacaine — 10 mg of a 5 mg/ml hyperbaric solution, intrathecally
  Other Names: Marcain; Local Anesthetic
Drug: Morphine — 200 µg of a 100 µg/ml solution, intrathecally
  Other Names: Intrathecal morphine
Drug: Lactated Ringer's solution — 25 ml/min intravenously
Drug: Ephedrine, continuous infusion — 37.5 mg/h intravenously
  Arms: Pharmacological
Drug: Ephedrine, bolus — 6.25 mg IV bolus prn.
  Hypotension defined according to study protocol for each arm.
Drug: Atropine — 0.1 mg/kg iv bolus prn
  Bradycardia defined as 50% drop in heart rate from baseline values.

SUMMARY:
The aim of this study is to compare two different therapeutic approaches to blood pressure reduction: pharmacological vs. non-pharmacological. The setting is that of patients undergoing scheduled Cesarean section under spinal anesthesia and suffering from aorta-caval compression syndrome, which causes a sudden drop in blood pressure.

DETAILED DESCRIPTION:
The supine hypotensive syndrome of pregnancy is induced by compression of the inferior caval vein by the enlarged uterus. It occurs in approximately 8% of pregnant women at term. More patients may develop an asymptomatic variety of this syndrome in the supine position. The hypotensive effect of spinal anesthesia per se may thus be aggravated in a significant number of term parturients. A preoperative supine stress test (SST) before elective cesarean section under spinal anesthesia has been shown to predict severe systolic hypotension with reasonable accuracy.

Different strategies have been proposed for the management of this complication; they can be divided into pharmacological and non-pharmacological ones.

According to pharmacological strategies, vasoactive drugs are used to treat hypotension induced by sympathetic efferent blockade following spinal anesthesia. To this end, α-agonist ephedrine is commonly considered the best choice because of its minimal impact on the fetoplacental circulation. However, excessive use of ephedrine may be detrimental to neonatal well-being because of its vasoconstrictor effect on fetoplacental circulation.

Non-pharmacological treatments may represent a valuable, safer alternative. According to many authors non-pharmacological treatments aimed at removing the cause of aorta-caval compression syndrome are to be preferred because more appropriate from an etiopathogenetic point of view. The use of a wedge-shaped cushion placed under the right hip is a well-known non-pharmacological strategy which allows the uterine left lateral displacement and, consequently, the removing of the compression from the inferior vena cava.

The aim of the present study is to compare, through the evaluation of neonatal well-being, the efficacy of these approaches to hypotension after spinal anesthesia for elective Caesarean section in parturients affected by aorto-caval compression.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal anesthesia for elective Cesarean section
* Patients in ASA Physical Status Class I or II
* Informed written consent to participation
* Positive Supine Stress Test

Exclusion Criteria:

* Any known fetal pathology
* Indication to general anesthesia
* Known allergy to any of the study drugs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Neonatal arterial base excess | <5 min from birth

SECONDARY OUTCOMES:
Neonatal arterial and venous pH, venous base excess | <5 min from birth
Apgar score | 1 and 5 minutes from birth
Maternal serum levels of cardiac troponin (baseline, immediate postsurgery, 6 and 12 hours after surgery) | Baseline and up to 12 h postoperatively
Incidence of maternal hypotension ( <20% baseline or mean arterial pressure <60 mmHg). | q5min from anesthesia to end of surgery
Incidence of maternal bradycardia (heart rate <30% of baseline or <60 beats per minute) | q5min from anesthesia to end of surgery
Peripheral arterial oxygen saturation: incidence of desaturation (SpO2 <92%) and mean values for each arm. | q5min from anesthesia to end of surgery
Administered atropine | from anesthesia to end of surgery
Amount of ephedrine administered (mg) | from anesthesia to end of surgery
Time between induction of anesthesia and skin incision
Time between skin incision and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fanelli, MD, Study Chair — Dept. of Anesthesiology and Critical Care Medicine, University of Parma, Italy; Andrea Cornini, MD, Study Director — UO II Anestesia, Rianimazione e Terapia Antalgica, Azienda Ospedaliero-Universitaria di Parma; Michele Zasa, MD, Principal Investigator — Dept. of Anesthesiology and Critical Care Medicine, University of Parma, Italy
Locations (1):
- University and Hospital of Parma (Azienda Ospedaliero-Universitaria di Parma), Parma, PR, Italy

REFERENCES:
- [Background] Kinsella SM, Lohmann G. Supine hypotensive syndrome. Obstet Gynecol. 1994 May;83(5 Pt 1):774-88. PMID 8164943
- [Background] Cyna AM, Andrew M, Emmett RS, Middleton P, Simmons SW. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD002251. doi: 10.1002/14651858.CD002251.pub2. PMID 17054153
- [Background] Kinsella SM, Norris MC. Advance prediction of hypotension at cesarean delivery under spinal anesthesia. Int J Obstet Anesth. 1996 Jan;5(1):3-7. doi: 10.1016/s0959-289x(96)80067-7. PMID 15321375
- [Background] Helwig JT, Parer JT, Kilpatrick SJ, Laros RK Jr. Umbilical cord blood acid-base state: what is normal? Am J Obstet Gynecol. 1996 Jun;174(6):1807-12; discussion 1812-4. doi: 10.1016/s0002-9378(96)70214-4. PMID 8678144